CLINICAL TRIAL: NCT00404703
Title: An Open Label Study of the Safety of First-line Treatment With Avastin in Combination With Cisplatin-gemcitabine or Carboplatin-paclitaxel in Patients With Advanced or Recurrent Squamous Non-small Cell Lung Cancer, Who Are Considered to be at High Risk of Pulmonary Haemorrhage
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Platinum-Based Chemotherapy in Patients With Advanced or Recurrent Squamous Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary (safety) endpoint reached
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO19734
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2008-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Platinum Compounds

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: Platinum-based chemotherapy

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 15mg iv on day 1 of each 3 week cycle
Drug: Platinum-based chemotherapy — As prescribed

SUMMARY:
This single arm study will assess the feasibility of using Avastin plus platinum-based chemotherapy (cisplatin-gemcitabine or carboplatin-paclitaxel) in patients with advanced or recurrent squamous non-small cell lung cancer who have not received prior chemotherapy. Patients will receive preventive radiation, followed by one cycle of chemotherapy alone and 5 cycles of chemotherapy in combination with Avastin (15mg/kg iv on day 1 of each 3 weekly cycle), followed by Avastin alone for a maximum total treatment period with Avastin of 12 months. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* documented squamous non-small cell lung cancer;
* stage IIIb with pleural or pericardial effusion, stage IV, or recurrent disease;
* suitable for platinum-based treatment as first line chemotherapy.

Exclusion Criteria:

* prior systemic anti-tumor therapy;
* prior radiotherapy for treatment of patient's current stage of disease;
* other primary tumors within last 5 years, except for controlled limited basal cell or squamous cancer of the skin, or cancer in situ of the cervix;
* major surgery, open biopsy or significant traumatic injury within 28 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Rate of grade >=3 Avastin-related pulmonary hemorrhage | After a maximum of 12 months treatment

SECONDARY OUTCOMES:
Overall response, duration of response, progression-free survival. | Event driven
AEs, laboratory parameters, coagulation parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- Australia (2):
  - Tugun
  - Wollongong
- Liège, Belgium
- Czechia (2):
  - Ostrava
  - Ústí nad Labem
- France (3):
  - Bobigny
  - Marseille
  - Nantes
- Hungary (2):
  - Székesfehérvár
  - Szombathely
- Israel (2):
  - Kfar Saba
  - Ramat Gan
- Poland (4):
  - Lublin
  - Poznan
  - Szczecin
  - Warsaw
- Russia (3):
  - Balashikha
  - Moscow
  - Saint Petersburg
- Spain (2):
  - Madrid
  - Seville
- Taiwan (4):
  - Kueishan
  - Taichung
  - Taipei
  - Taoyuan District